CLINICAL TRIAL: NCT03357458
Title: Parent-child Interactions, Child Developmental Health, and Health System Costs at 6 Months Corrected Age: Effectiveness of a Cluster Randomized Controlled Trial of Family Integrated Care in Level II NICUs
Brief Title: Parent-child Interactions, Child Developmental Health, and Health System Costs at 6 Months Corrected Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ACHRI FICare 6mth
Record Dates: First submitted 2017-10-23; First posted 2017-11-30 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Preterm Birth; Prematurity; Infant,Premature; Infant Development; Child Development; Parent-Child Relations; Mental Health Wellness 1
Keywords: Family Integrated Care; Parenting education; Nursing; Cost effectiveness; Patient engagement; Randomized controlled trial; Neonatal intensive care unit
MeSH Terms: conditions — Premature Birth; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Integrated Care (Experimental): Study participants receive FICare, a dynamic psycho-educational intervention, while their infant(s) was/were admitted to a Level II NICU.
  Interventions: Behavioral: Family Integrated Care
- FICare Control Group (No Intervention): Study participants received standard care while their infant(s) was/were admitted to a Level II NICU.

INTERVENTIONS:
Behavioral: Family Integrated Care — FICare is a dynamic psycho-educational intervention. The goal of FICare is a change in culture and practice that permits, encourages and supports parents in their parenting role while their infant is receiving health care in a Level II NICU. Underpinned by adult learning and change theories, FICare empowers parents to build their knowledge, skill and confidence so that the family is well-prepared to care for their infant long before discharge.
  Arms: Family Integrated Care

SUMMARY:
The aim of this novel health services research proposal is to assess the longer-term outcomes, to 6 months corrected age, of an adapted Family Integrated Care (FICare) model of care for moderate and late preterm infants admitted to a Level II neonatal intensive care unit (NICU).

This follow-up study will enroll infants at 6 months CA (± 1 month) recruited to the original FICare randomized controlled trial (clinicaltrials.gov ID: NCT02879799) from four level II NICU sites; two intervention and two control.

DETAILED DESCRIPTION:
The aim of this novel health services research proposal is to assess the longer-term outcomes, to 6 months corrected age, of Family Integrated Care (FICare) for moderate and late preterm infants admitted to a Level II neonatal intensive care unit (NICU). FICare is a psycho-educational intervention that empowers parents (mothers and fathers) to sequentially build their knowledge, skill, and confidence so the family is well-prepared to care for their preterm infant before discharge. FICare is dynamic, whereby parents and healthcare providers openly and mutually negotiate equitable caregiving roles during the infant's NICU stay. Parents are educated and coached to provide routine non-medical care. Healthcare providers continue to provide medical and technical care, such as intravenous medications and procedures, legal documentation, and professional support for families. Using a cluster randomized controlled trial (cRCT), our team is evaluating FICare in all 10 Level II NICUs in Alberta (5 intervention, 5 control sites; stratified by hospital size) with follow-up of infant development and costs at age 2 months corrected age (CA). Unless otherwise indicated, infant ages are corrected for prematurity. For the cRCT, we hypothesized that FICare would reduce length of NICU stay by 10%, reduce infant morbidities (e.g., nosocomial infections, respiratory support, feeding problems), increase breast-milk feeding, reduce maternal psychological distress, and reduce costs to the health care system and families. Maternal and infant data are currently being collected (1) shortly after admission to the NICU (baseline), (2) shortly before discharge from NICU (outcome), and (3) at 2 months CA (follow-up). At 2 months CA, our team will evaluate outcomes related to infant global development and maternal psychosocial distress. A follow-up study at 6 months CA will provide evidence of the sustainability of any effects, upon which to inform policy decisions about full-scale implementation of FICare in Level II NICUs.

There is currently no standardized timeline for follow-up of infants born prematurely. Follow-up at 6 months CA is appropriate as the utility of assessing development in preterm infants is questionable prior to this age, and evidence suggests that inter-individual variability in child development increases after 12 months. After 12 months, it becomes more difficult to capture parent-child interactions and environmental factors may exert a stronger influence on infant development, potentially diluting the ability to directly measure the effect of FICare.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants born between 32 weeks and zero days and 34 weeks and 6 days gestation who enrolled in the FICare Alberta cluster controlled trial (cRCT) at one of four of the ten Level II NICU sites. The FICare cRCT enrolled mothers of any age who have decision making capacity; mothers who are able to speak, read and understand English well enough to provide informed consent, and complete surveys online or via telephone.

Exclusion Criteria:

* The FICare Alberta Level II NICU cRCT excluded mothers whose infants have serious congenital or chromosomal anomalies that require surgery, or are receiving palliative care; mothers who are not able to communicate in English; mothers with complex social issues.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Maternal-Child Interactions | At 6-months corrected age
  We will measure maternal-child interactions using the Parent-child interaction Teaching Scale (PCITS) to code video-taped structured play sessions of mothers with their infants. The PCITS is the most widely used macro-level, binary observational measure of the presence or absence of dyadic behaviours. The parent total (50 items; possible score of 50) is the sum of subscales: Sensitivity to Cues, Response to Distress, Social-Emotional Growth Fostering, and Cognitive Growth Fostering. The child total (23 items; possible score of 23) is the sum of subscales: Responsiveness to Caregiver and Clarity of Cues. Higher scores indicate more optimal interactions. It has been validated with preterm infants.

SECONDARY OUTCOMES:
Infant global development | At 6-months corrected age
  Ages and Stages Questionnaire, 3rd edition: developmental screening instrument consists of 21 age-appropriate (1 to 66 months of age) questionnaires, with 30 items each. Assesses development in 5 domains: communication, gross motor, fine motor, problem-solving, and personal-social, each consisting of 6 items. Responses for each item receive a score of 0, 5, or 10 points. Item scores are summed for a total score with a possible range of 0 to 60 for all domains. Higher scores indicate more optimal child development. Based on empirically derived cut-offs, each domain total score is classified as (a) appropriate development, (b) monitoring zone (≥1 and < 2 standard deviations below the mean), and (c) need for referral (2 standard deviations below the mean). The ASQ-3 has strong psychometric properties, including high sensitivity (0.86) and specificity (0.85), and has been evaluated and recommended as an effective screener of global development in moderate and late preterm infants
Infant social and emotional development | At 6-months corrected age
  Ages and Stages Questionnaire:Social-Emotional, 2nd edition: Screening instrument focused specifically on the social-emotional development of infants and young children, consisting of 9 age-appropriate (1 to 72 months of age) questionnaires. Scale at 18-months consists of 31 items, each receives a score of 0, 5, 10, or 15 points. Item scores are summed for a total score with a possible range of 0 to 465 (score of 105 represents 90th percentile). Lower total scores indicate more optimal social-emotional development. Based on empirically derived cut-offs, the total score is classified as (a) appropriate social-emotional development (below 65th percentile), (b) monitoring zone (between 65th percentile and referral cut-off), and (c) need for referral (above referral cut-off; around 80th percentile, depending on age interval). Test-retest reliability (0.89) and internal consistency reliability (0.84) are high, as are overall sensitivity (81%) and specificity (84%).
Maternal-reported infant sleep | At 6-months corrected age
  Extended Brief Infant Sleep Questionnaire (EBISQ): As the EBISQ is not a psychometric scale, no composite score is calculated, nor are there sub-scale. The scale contains 32 items capturing information on infant sleep patterns, sleep ecology, and caregiver perceptions; response categories include numerical (time, frequency count of night wakings), categorical (sleep location, bedtime activities) and ordinal rankings (how much of a problem is your baby's sleep? A large problem, a small problem, or no problem). No numerical values are assigned to items with ordinal or categorical answers. The EBISQ has been validated against actigraphy and daily-logs and its sensitivity in documenting expected developmental changes in infant sleep and the effects of environmental factors has been established.
Maternal parenting self-efficacy | At 6-months corrected age
  Perceived Maternal Parenting Self-Efficacy Scale: A 20 item self-report measure of maternal parenting self-efficacy, scored on a 4-point Likert scale. The total score is calculated as a sum of responses to all 20 questions. Mothers can score between 20 - 80 overall, where the higher the score the higher the self-efficacy. Four subscales reflect different aspects of parenting, however; there are no cut-off scores.
Breastfeeding rates | At 6-months corrected age
  Breastfeeding questionnaire: a non-pscyhometric questionnaire will evaluate breastfeeding rates with questions asking if participants are breastfeeding, frequency of breastfeeding, and if participants are not breastfeeding, we ask infant's age at weaning and why breastfeeding was stopped.
Number of emergency room visits | At 6-months corrected age
  Provincial healthcare administrative databases
Number of re-admissions to hospital | At 6-months corrected age
  Provincial healthcare administrative databases
Number of unplanned visits to physician or other provider | At 6-months corrected age
  Provincial healthcare administrative databases
Number of antibiotic prescriptions | At 6-months corrected age
  This data will be collected in two ways: 1) maternal self-report as part of a study questionnaire, and 2) from the patient chart as collected by Alberta Health Services (AHS), the provincial healthcare provider in Alberta, Canada. A data disclosure agreement has been executed such that AHS Analysts with the Analytics, Data Integration, Measurement & Reporting (DIMR) team will link FICare data with fields related to the number antibiotic prescriptions in AHS data holdings. The specific variables related to this outcome will be selected for and identified in consultation with AHS Analysts who have extensive knowledge of their metadata.
Direct industry costs (hospital costs, excluding housekeeping, maintenance, planning and physician times). | At 6-months corrected age
  Provincial healthcare administrative databases
Parenting stress | At 6-months corrected age
  Parenting Stress Index - Short Form - 4th edition (PSI-SF-4): A 36-item scale, captures general parenting stress and three subscales of Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Responses 1, 2, 3, 7, 8, 9 and 11 are summed for Defensive Responding. Subscale scores are calculated by summing response items 1-12 for Parental Distress, items 13 - 24 for Parent-Child Dysfunctional Interaction, and items 25 - 36 for Difficult Child. Total Stress score is calculated by summing the raw scores of the subscales. Raw scores are converted to T scores and percentiles. Normal range for scores is within the 16th to 84th percentiles. Scores in the 85th to 89th percentile are considered high, and scores in the 90th percentile or higher are considered clinically significant.
State Anxiety | At 6-months corrected age
  State-Trait Anxiety Inventory (STAI): Two sub-scales: 1) long-standing quality of trait anxiety (20 items), and 2) the temporary condition of state anxiety (20 items). Items are rated on a 4-point scale. Item scores are added to obtain subtest total scores. Scoring is reversed for anxiety-absent items (19/40 items). Range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the state anxiety scale. Normative values are available in the manual. Trait anxiety was collected previously in the FICare cRCT (NCT02879799) therefore, only state anxiety will be collected at 6 months.
Postnatal depression risk | At 6-months corrected age
  Edinburgh Postnatal Risk Depression (EPDS) scale: A 10 item, 4-point Likert scale, self-report measure of postnatal depression. The total score is calculated as a sum of responses to all 10 questions. Questions 1, 2 and 4 are reverse scored. The range of possible scores are: 1) 0-9; indicates presence of some symptoms of distress that may be short-lived and less likely to interfere with day to day ability to function, 2) 10 - 12; indicate presence of symptoms of distress that may be discomforting, and 3) 13+; requires further assessment and appropriate management as likelihood of depression is high. Referral to professional supports may be necessary. Any woman scoring 1+ on item 10 requires further evaluation to ensure her own safety and that of her baby/babies.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Discussions are underway to draft a data deposition agreement with Secondary Analyses to Generate Evidence (SAGE).